CLINICAL TRIAL: NCT00846261
Title: The Infected Bone Nonunion and Soft Tissue Defect of Long Bone Treated Simultaneously With Ilizarov Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Department of Orthopedics, 2nd Affiliated Hospital, School of Medicine,, Zhejiang University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Z2-001
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Trauma; Orthopedic Surgery Complications
Keywords: infected; Ilizarov
MeSH Terms: conditions — Wounds and Injuries | interventions — Ilizarov Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ilzarov (Experimental)
  Interventions: Device: Use it to treatment bone nonunion (Ilzarov)

INTERVENTIONS:
Device: Use it to treatment bone nonunion (Ilzarov) — Detect the variation of limb lengthening
  Other Names: Ilizarov; Trauma

SUMMARY:
In this retrospective study, the investigators evaluated the clinical and functional results of infected nonunion of the long bone with soft-tissue defects treated simultaneously with Ilizarov technique combining open dressing change in 22 patients. The investigators wanted to find out whether that the internal bone transport with external fixator combining open dressing change is a valuable method to treatment for those patients with infected bone nonunion and poor condition of the soft tissue such as sinus, skin defect.

DETAILED DESCRIPTION:
From January 2002 to now, totally 22 patients (18 males, 4 females) were underwent internal bone transport for infected nonunion in the long bone with soft-tissue defects. The mean age of the patients was 36.5 years (range, 19 to 57). The infected nonunion occurred on the femur in 1 patients, the tibia in 21 patients. The hybrid mono-lateral limb reconstruction external fixator was used, combined with bone transport. The results were evaluated by the classification of the Association for the Study and Application of the Method of Ilizarov (ASAMI) which divided into bone and functional categories

ELIGIBILITY:
Inclusion Criteria:

* Patients with infected nonunion of long bone with soft tissue defects or sinus, without systemic illness that could affect their immunologic status (e.g., AIDS, diabetes mellitus, liver cirrhosis).

Exclusion Criteria:

* Patient noncooperation and an age of less than 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-01; Primary Completion 2006-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Achive wounds close and bone union | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zheng, doctor, Study Director — Department of Orthopedics, 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China